CLINICAL TRIAL: NCT02949544
Title: Water Immersion and Water-based Exercise in Patients With Chronic Stable Heart Failure: A Pilot Study
Brief Title: Water Immersion in Chronic Stable Heart Failure
Acronym: IMMERSE-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R1996
Record Dates: First submitted 2016-10-13; First posted 2016-10-31 (Estimated); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Masking Description: open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- water immersion (Other): patients with heart failure will be immersed to the neck for 15 minutes
  Interventions: Other: water immersion

INTERVENTIONS:
Other: water immersion — warm water immersion

SUMMARY:
This study aims to investigate the effects of water immersion and exercise on heart function and blood flow in patients with chronic stable heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* Established diagnosis of heart failure with NTpro BNP >100

Exclusion Criteria:

* Uncontrolled or severe heart failure, defined by NYHA class IV symptoms (breathlessness at rest)
* Severe fluid overload characterised as more than minimal pitting oedema of the ankles only
* Presence of haemodynamically significant valvular heart disease in the opinion of the investigator
* Haemoglobin <125 g/L
* Weight >120 kilograms
* Requiring long term oxygen supplementation in the community
* Hospitalisation for any cause within the last 6 weeks, that in the opinion of the investigator would affect the patients wellbeing in this study
* Unstable or severe stable angina that requires three or more antianginals
* Patients known to have disease causing immunocompromise such as HIV infection or undergoing chemotherapy
* Patients with active infection
* Dialysis patients
* Uncontrolled seizures; patients in whom the pool environment may trigger seizures, new diagnosis of epilepsy
* Insulin treated diabetic patients with hypoglycaemic episodes in the last 3 months.
* Pregnant women
* Central venous lines which are not tunnelled and are exposed superficially.
* Open access ports to lungs including tracheotomy sites
* Ventilation tubes for ears
* Nasogastric or gastrostomy tube in situ
* Presence of colostomy, ileostomy or urostomy.
* Presence of open, macerated, infected or non-intact skin or oedema with leakage of serous fluid.
* Skin condition such as severe eczema or psoriasis
* Any surgery or invasive devices fitted within the last 4 weeks
* Any form of mobility impairment requiring mobility aids (e.g. stick or wheelchair) or rendering patient unable to perform gentle exercises, including recent injury or trauma
* History of chlorine sensitivity
* Urinary or faecal incontinence
* Hydrophobia
* Unable to give consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2016-11-22 (Actual); Primary Completion 2017-04-04 (Actual); Study Completion 2017-04-04 (Actual)

PRIMARY OUTCOMES:
Cardiac output | 15 minutes of water immersion

SECONDARY OUTCOMES:
Heart rate (beats/minute) | 15 minutes of water immersion
Blood pressure (mmHg) | 15 minutes of water immersion
systemic vascular resistance (dyn·s/cm5) | 15 minutes of water immersion
Stroke volume (millilitres) | 15 minutes of water immersion
Jugular venous pressure (not raised, raised 1-4cm, raised to earlobes, undetectable) | 15 minutes of water immersion
BORG dyspnoea score (score between 1-10) | 15 minutes of water immersion
cardiac output (milliliters/minute) | 3 minutes of exercise in water
N-terminal pro b-type natriuretic peptide (ng/L) | 10 mins after water immersion
Left ventricular end systolic diameter (mm) | 15 minutes of water immersion
Left ventricular end diastolic diameters (mm) | 15 minutes of water immersion

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Clark, Principal Investigator — Castle Hill Hospital
Locations (1):
- Castle Hill Hospital, Cottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Shah P, Pellicori P, Kallvikbacka-Bennett A, Zhang J, Pan D, Clark AL. Warm water immersion in patients with chronic heart failure: a pilot study : Shah immerse: HF. Clin Res Cardiol. 2019 May;108(5):468-476. doi: 10.1007/s00392-018-1376-2. Epub 2018 Sep 28. PMID 30267153
- See also: Full PDF Original Paper — https://link.springer.com/content/pdf/10.1007%2Fs00392-018-1376-2.pdf